CLINICAL TRIAL: NCT04134065
Title: the Effect of Target-oriented Vitamin D Treatment in Refractory Crohn's Disease
Brief Title: the Effect of Vitamin D in Crohn's Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing University School of Medicine (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Lei Zheng, Clinical Professor, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJUSM
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Vitamin D Deficiency; Crohn Disease
Keywords: Vitamin D; Crohn Disease; recurrence
MeSH Terms: conditions — Vitamin D Deficiency; Crohn Disease; Recurrence | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The physical properties such as appearance, size, color, dosage form, weight, taste and odor of placebo should be as much as possible as the test drug, but should not contain the Vitamin D (such as tablets containing lactose).
  Interventions: Drug: Placebo oral capsule
- Vitamin D group (Experimental): Liquid cholecalciferol supplementation (OsteVit DTM, Key Pharmaceuticals, Macquarie Park, NSW, Australia), supplied in 50 mL bottles (5000 units in 1 mL)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — patients with refractory Crohn disease and a serum 25(OH)D concentration <75 nmol/L were prescribed oral liquid vitamin D supplementation over 12 weeks using a specific protocol with dose adjusted 4-weekly to aim for a target level of 100e125 nmol/L.
  Other Names: VD
  Arms: Vitamin D group
Drug: Placebo oral capsule — the capsule contain nothing
  Other Names: Placebo
  Arms: Control group

SUMMARY:
To evaluate the efficacy and safety of 12-week goal-directed therapy in the treatment of refractory inflammatory patients, and to initially explore treatment options. Patients with potential risk factors for recurrence after surgery for Crohn's disease and a serum 25(OH)D concentration <75 nmol/L were prescribed oral liquid vitamin D supplementation over 12 weeks using a specific protocol with dose adjusted 4-weekly to aim for a target level of 100-125 nmol/L.

DETAILED DESCRIPTION:
The patients received oral liquid cholecalciferol supplementation (OsteVit DTM, Key Pharmaceuticals, Macquarie Park, NSW, Australia), supplied in 50 mL bottles (5000 units in 1 mL). A target 25(OH)D of 100-125 nmol/L was planned and the dose titrated 4-weekly.

Patients were evaluated at week 0 (screening visit), then 2- weekly until week 12, and at a follow-up visit at week 16. Key study endpoints were change in total 25(OH)D and attainment of level of 100e125 nmol/L. Intestinal inflammation was assessed via clinical disease activity (CDAI), faecal calprotectin (Calprotectin ELISA, Buhlmann, Basel, Switzerland), and circulating inflammatory markers (platelet count, serum albumin and C- reactive protein). Safety was assessed by direct questioning and 24- h urinary calcium excretion . Compliance was checked by dosing diaries completed by patients and measuring remaining cholecalciferol in bottles of the study drug.

Statistical analyses were performed using SPSS v20 (IBM Corporation, 2011) and GraphPad Prism v5.04 (Graphpad software, 2010). Dependent and independent samples t-tests, analysis of variance (ANOVA) and KruskaleWallis tests were used where appropriate. Associations with rise in 25(OH)D were examined by bivariate correlations. A p-value of 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Crohn's Disease
2. Must be able to swallow tablets
3. Have certain factors increase the risk of surgery in CD. include:

   * current smoking
   * fistulizing and stricturing disease behaviour
   * early steroid use (medical need for steroids for treatment of first flare)
   * disease in the end of the small bowel (i.e. ileum)
   * disease in the middle part of the small bowel (i.e. jejunum), and
   * young age at the time of the diagnosis.

Exclusion Criteria:

1. Other serious gastrointestinal diseases
2. pregnancy
3. hypercalcemia
4. hyperparathyroidism
5. chronic kidney disease and cardiovascular disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical disease activity | up to one year
  CDAI score
Fecal calprotectin | up to one year
  Calprotectin is a calcium-containing protein derived from neutrophils and macrophages. Its expression is tissue or cell specific and can be used as a marker for activation of acute inflammatory cells.
C-reactive protein | up to one year
  circulating inflammatory markers
Discomportant complaint | up to one year
  Incidence of Treatment Adverse Events
24-hour urinary calcium | up to one year
  Determination of calcium in urine for 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yousheng Li, Doctor, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg M, Rosella O, Rosella G, Wu Y, Lubel JS, Gibson PR. Evaluation of a 12-week targeted vitamin D supplementation regimen in patients with active inflammatory bowel disease. Clin Nutr. 2018 Aug;37(4):1375-1382. doi: 10.1016/j.clnu.2017.06.011. Epub 2017 Jun 15. PMID 28651829